CLINICAL TRIAL: NCT04973124
Title: Analyzing the Neuroprotective Effect of Dexmedetomidine in Terms of Preserving Brain Functional Connectivity in Elderly Patients After Major Surgery
Brief Title: The Neuroprotective Effect of Dexmedetomidine Preserving Brain Functional Connectivity in Elderly Patients
Acronym: DEXPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200618004
Record Dates: First submitted 2021-06-24; First posted 2021-07-22 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2024-11

CONDITIONS: Anesthesia; Dexmedetomidine; Aging
Keywords: Aged; Dexmedetomidine; Anesthesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to any of the groups: Control Group and DEX Group
Who Masked: Participant, Care Provider
Masking Description: Each participant will be assigned an identifier that the research team will use from enrollment to follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SEVODEX Group (Active Comparator): The SEVODEX group will receive intraoperative dexmedetomidine at a fixed infusion rate of 0.25 mcg/kg/h
  Interventions: Drug: Dexmedetomidine
- SEVO Group (Placebo Comparator): The SEVO group will not receive dexmedetomidine during surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — These participants will receive intraoperative dexmedetomidine.
  Other Names: Sevoflorane
  Arms: SEVODEX Group
Drug: Placebo — These participants will not receive intraoperative dexmedetomidine.
  Arms: SEVO Group

SUMMARY:
Older patients are more prone to adverse cognitive outcomes such as postoperative delirium (POD) and postoperative cognitive dysfunction (POCD). Both conditions are associated with an increased risk of death, functional decline, and health care costs. The presence of pro-inflammatory cytokines in the central nervous system has detrimental effects on the regulation of neurotransmitter signaling in different areas of the brain, especially the hippocampus, ultimately resulting in neuronal dysfunction and cognitive decline. Neuroimaging studies have provided important information on the structural and functional networks involved in the pathogenesis of POD and POCD. Strong evidence has shown a decrease in the integrity of the default mode network (DMN), along a continuum from normal aging to mild cognitive impairment and Alzheimer's disease. Dexmedetomidine is a highly selective alpha-2 adrenergic agonist with sedative and analgesic properties but minimal respiratory effects. Several studies have shown that dexmedetomidine reduces serum pro-inflammatory cytokines and POCD. The expected results are to analyze the change in the integrity of the DMN from the preoperative period to the first weeks after discharge given by the two anesthetic strategies (SEVO vs SEVODEX). In addition, it seeks to evaluate (1) Changes in the integrity of the DMN at 3 months. (2) Modulation of structural changes in white matter integrity as measured by DTI. (3) Patient performance in specific cognitive function tests and serum inflammation biomarkers between the pre- and postoperative period. For the analysis, the Generalized Linear Model (GLM) will be used, in which the integrity of the DMN is the dependent variable. As predictors will use the anesthetic groups (SEVO and SEVODEX) and the measurement time (preoperative, 1 to 3 weeks after discharge and 3 months later as levels). With this work we aim to provide a mechanistic explanation of the observed neuroprotective effects of dexmedetomidine in anesthesia protocols for elderly patients. Furthermore, this work will possibly promote functional connectivity as a possible clinical biomarker of cognitive impairment in this vulnerable population.

DETAILED DESCRIPTION:
Cognitive impairment after anesthesia in older patients The average age of the world population is rapidly increasing as is the number of elderly patients who undergo surgery. According to projections of the last census, the Chilean population is also undergoing a process of demographic ageing. Elder patients are more prone to adverse cognitive outcomes such as post-operative delirium (POD) and postoperative cognitive dysfunction (POCD). The observed overall incidence of POD and POCD is 40% and 10% respectively and both can represent transient or permanent brain damage. Both conditions are associated with an increased risk of death, functional decline, and health care costs. POD is an acute and transient condition that occurs during the first few days after surgery. In contrast, POCD manifests with more subtle deficits in memory, attention, and cognition over a much longer period of time (months to years). Even though the increase in age and the degree of frailty are well known risk factors for adverse postoperative cognitive outcomes, the etiology of these conditions remains poorly understood and most likely involves a combination of patient, surgical, and anesthetic factors.

Surgical trauma and inflammatory response Several studies in animals and humans have shown that surgical trauma triggers immune and inflammatory responses that can potentially generate neuroinflammation and degeneration. Neuroinflammation is a localized inflammation occurring in both the peripheral and central nervous system in response to trauma, neurodegeneration, bacterial or viral infection, autoimmunity and toxins. The pathogenesis of surgery-induced neuroinflammation involve the release of biomolecules known as damage-associated molecular patterns (DAMPs) such as the high molecular group box 1 protein (HMGB1). The various DAMPs molecules released activate nuclear factor-kappa B (NF-κB) signaling pathways in bone marrow derived monocytes20. The activated monocytes increase the activity and expression of cyclooxygenase 2 isozyme (COX-2), expression of pro-inﬂammatory cytokines interleukin-1 beta (IL-1β), interleukin 6 (IL-6), and tumor necrosis factor alpha (TNFα). These pro-inﬂammatory cytokines promote further release of HMGB1 from injured cells, further activation of monocytes, and finally disruption of the blood brain barrier allowing pro-inﬂammatory mediators to enter the central nervous system.

Several studies have shown that the magnitude of postoperative cognitive impairment is strongly associated with the levels of pain and inflammation. Major surgeries, like cardiac surgery and major orthopedic surgery, have been associated with POCD in up to 50% of patients. Regarding memory formation and brain cognitive processes, the presence of pro-inﬂammatory cytokines in the central nervous system have detrimental effects on the regulation of neurotransmitter signaling in different brain areas, especially the hippocampus, ultimately resulting in neuronal dysfunction and cognitive impairment. For example, the hippocampus is readily affected by pro-inﬂammatory factors, which break the α-amino-3-hydroxy-5-methyl-4-isoxazolepropionic acid (AMPA)-to- N-Methyl-d-aspartic acid or N-Methyl-d-aspartate (NMDA) balance in glutamatergic synapsis, disrupting the process of long-term potentiation, and thus the ability to form memories. Additionally, HMGB1 produced in the brain increases the influx of glutamate in hippocampal neurons, which ultimately results in glutamate toxicity, neuronal death and cognitive impairment.

Anesthetic neurotoxicity Anesthetics induced neurotoxicity has become an area of great concern in recent decades due to numerous studies showing anaesthetics may promote neuroapoptosis in immature brains of animals. Although, general anesthetics are normally considered safe in adults, several studies suggest that anesthetic exposure is associated with postoperative cognitive dysfunction in adult patients. Most used inhaled general anesthetics (isoflurane, sevoflurane and desflurane) are highly lipid-soluble and can rapidly access the brain in high concentrations. Since they act on many receptors, such as γ-aminobutyric acid (GABA) and NMDA receptors, second messenger systems, enzymes, and even cytoskeletal components, it is not surprising that they might be involved in neurodegenerative changes in vulnerable populations, especially after high concentrations and long exposure times. There is strong evidence in animals to support that exposure to anesthetics can induce dose-dependent neurotoxicity. Cellular degeneration from isoflurane exposure have shown to result in altered white matter integrity indicating damage in fiber tracts, leading to the development of neurological and cognitive deficits. In addition, volatile anesthetics have been shown to increase concentrations of the β-amyloid protein and can lead to hyperphosphorylation of the tau protein, changes that are paramount in the cytotoxicity of Alzheimer's disease. Studies using in vitro models have provided consistent evidence that volatile general anesthetics suppress transmission in different types of synapses, altering neuronal network excitability.

Dexmedetomidine neuroprotection Dexmedetomidine is a highly selective alfa-2 adrenergic agonist with sedative and analgesic properties but minimal respiratory effects. Dexmedetomidine produces its sedative effects by acting at the locus coeruleus, analogous to the natural induction of sleep, and independent of NMDA or GABAA receptors. In intensive care units, dexmedetomidine's anti-inflammatory, organ-protective, and sympatholytic effects have been associated to better outcomes when compared to benzodiazepine sedative regimes. A recent study in septic patients showed that individuals receiving dexmedetomidine had more days free of brain dysfunction and were less likely to die than those that received lorazepam sedation. There is also growing evidence of dexmedetomidine organ protective properties in ischemia reperfusion, inflammation, and traumatic brain injury models. A randomized control trial reported a 60% reduction of POD after an infusion of dexmedetomidine. Another randomized controlled trial showed improved cognitive function and quality of life in 3-year survivors, as well as increasing survival up to 2-years after a low-dose dexmedetomidine infusion in non-cardiac surgery. In a recent meta-analysis, dexmedetomidine administration showed an overall 40% reduction in the risk of POCD.

Although the underlying neuroprotective mechanisms of dexmedetomidine are not clear, several mechanisms have been proposed. In animal models, dexmedetomidine has been shown to reduce the severity of neuroinflammation, neuro apoptosis, expression of IL-1β, IL-6, TNF-α and TLR-4, as well as the reduction of astrocyte and microglial activation. It also has been shown that it promotes the recovery of neurogenesis in aged mouse in a model of postoperative cognitive dysfunction. Other researchers have suggested that the protective effect may be due to an inhibitory effect in the gap junctions, which are involved in the integrity of the brain blood barrier. In addition, dexmedetomidine administration has been shown to reduce sevoflurane-induced apoptosis in several cortical and subcortical brain regions of neonatal rats. Human studies have shown that dexmedetomidine reduces serum pro-inﬂammatory cytokines and POCD compared to saline on postoperative day 1 in patients undergoing laparoscopic cholecystectomy. A recent study showed a correlation between the level of reduction of pro-inﬂammatory cytokines and POCD on postoperative day 1, suggesting a link between cytokine levels and the severity of cognitive dysfunction. The protective effects of dexmedetomidine from cognitive dysfunction in surgical contexts is relatively well established. The main proposed molecular mechanism of action is believed to be due to a reduction of neuroinflammation. However, in terms of brain activity patterns, the questions of how volatile anesthetics are increasing the risk of cognitive dysfunction, and how dexmedetomidine protects against these risks remains largely unknown.

Magnetic Resonance Imaging Recent advances in magnetic resonance imaging (MRI) methods bring new opportunities to study neuronal activity and neuroplastic changes of the human brain. In broad terms, MRI analysis can be separated into structural and functional methods. In terms of brain structure, a previous study found that patients with white matter abnormalities in the cerebellum, hippocampi, thalami and the anterior brain, observed using diffusion tensor imaging (DTI) prior to surgery, were associated with a higher incidence and severity of delirium. In a follow-up study of the same patients performed one year after surgery, the authors found that white matter abnormalities of the frontal, parietal, and temporal lobes were associated with delirium severity Although, the evidence is still scarce and the results of previous studies have shown inconsistencies between MRI structural markers and clinical findings, the possibility of being able to observe direct biomarkers of cerebrovascular and neurodegenerative features of brain damage appear as a valuable approach to improve our understanding of the underlying mechanisms behind POD and POCD.

Functional connectivity and the Default mode network In addition to structural analysis, MRI allows for the study of the dynamics of the functioning brain. At rest, specific brain areas show coherent activation, measured as the correlation of their Blood Oxygen-Level Dependent (BOLD) signal. The most prominent of these networks is the Default Mode Network (DMN), which arises spontaneously in normally functioning brains when at rest. The DMN comprises a collection of brain regions including the medial prefrontal cortex (mPFC), posterior cingulate cortex (PCC), precuneus, anterior cingulate cortex (ACC), parietal cortex, and the hippocampus. This network is particularly relevant for aging and dementia since DMN structures are vulnerable to atrophy, deposition of the amyloid protein, and generally show a reduced glucose metabolism. Neuroimaging studies have provided important information about the functional networks involved in POD and POCD pathogenesis.

Solid evidence has shown a decreased in the integrity of the DMN (reduced functional connectivity) along a continuum from normal aging to mild cognitive impairment and to Alzheimer's disease. However, in the context of post-operative cognitive decline, previous neuroimaging studies have focused on finding patient's features as predictors of POD and POCD, leaving aside the possible effect that the anesthesia technique could have on the surgery-induced disruption of the DMN and its link to cognitive impairment. Here we propose to study the neuroprotective effect of dexmedetomidine in terms of neuroinflammation but also in terms of the preservation of the integrity of functional and structural connectivity in a brain network known to be affected in patients with cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* ASA I, II or III.
* Body mass index (BMI) <35 kg/m2.
* Scheduled at least 6 days prior to surgery to allow adequate time for the baseline assessment.
* Planned admission to the hospital for at least 2 days.

Exclusion Criteria:

* Active delirium diagnosed with the Confusion Assessment Method (CAM).
* Mild cognitive impairment or dementia diagnosed with the Spanish-language version of the Montreal Cognitive Assessment MoCA-S1-2 score (score <20 points).
* In case the patient cannot answer the MoCA test, the instrument AD8-Ch will be applied.
* Hospitalization within 3 months prior to enrollment to minimize risk of recent delirium history.
* Severely frail condition defined with the Clinical Frailty Scale (CFS ≥7).
* Inability to perform cognitive tests due to legal blindness or severe deafness
* History of schizophrenia or psychosis.
* Harmful alcohol use or alcohol dependence (AUDIT score ≥16 considering the standard drink equivalent determined by MINSAL).
* History of benzodiazepines or marihuana consumption (more than 3 days per week).
* Unable to pass assessment for capacity to provide informed consent.
* Claustrophobia.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Reduction of the alteration of the NDM due to the effect of dexmedetomidine associated with sevoflouran in elderly patients under general anesthesia | f-MRI before surgery (t0), f-MRI two to four weeks post discharge (t1), Three months post discharge (t2)
  To assess the effect of the administration of dexmedetomidine, together with sevoflurane, in reducing the disruption of the default mode network (DMN) after surgery in elderly patients through functional magnetic resonance imaging( f-MRI)of the brain.

SECONDARY OUTCOMES:
The relationship among the indicators of systemic inflammation and Cognition | Pre and postoperative levels of IL-6, TNFα and pre and postoperative score of the MoCa test up to 3 month.
  To analyze the relationship among the indicators of systemic inflammation IL-6 pg/dL and TNFα pg/dL and the score of the cognitive test (score MoCA-S1-2 test) with changes in the Surgery-induced functional connectivity in two anesthetic conditions, association among the variables depending on the observed normality, using the Pearson correlation or the Spearman correlation
The relationship among the indicators of systemic inflammation and Delirum | Pre and postoperative levels of IL-6, TNFα and pre and postoperative score of CAM up to 7 days.
  To analyze the relationship among the indicators of systemic inflammation (IL-6 and TNFα) and the Delirum (screening Confusion Assessment Method -CAM) with changes in the surgery-induced functional connectivity in two anesthetic conditions, association among the variables depending on the observed normality, using the Wilcoxon-Mann-Whitney or t-test.
The relationship among the indicators of systemic inflammation and frailty . | Pre and postoperative levels of IL-6, TNFα and pre and postoperative score of frail scale up to 7 days.
  To analyze the relationship among the indicators of systemic inflammation (IL-6 and TNFα) and the score of the cognitive test (score MoCA-S1-2 test) and frailty (FRAIL scale) with changes in the surgery-induced functional connectivity in two anesthetic conditions, association among the variables depending on the observed normality, using the Wilcoxon-Mann-Whitney or t-test
The association between poor cognitive outcomes and potential markers brain injury. | Pre Operative score MoCa test, CAM and f-MRI (t0) and Post Operative score MoCa test, CAM and f-MRI (t2) up to 3 months.
  To explore the association between poor cognitive outcomes (measured by MoCa Test and CAM) and potential markers of magnetic resonance brain injury (functional and structural) measured by f-MRI. Association among the variables depending on the observed normality, using the Wilcoxon-Mann-Whitney or t-test
The association between postoperative neuroinflammation and images of brain structure | Post operative IL-6, TNFα and f-MRI (t2) up to 3 months.
  Compare the magnitude of postoperative neuroinflammation (measured by IL-6 pg/dL and TNFα pg/dL) and post operative MRI results (measured by structural f-MRI) up to 3 months using the ANOVA-test or Mann-Whitney U.

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Cortinez, MD, Principal Investigator — Titular Profesor
Locations (1):
- Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown EN, Purdon PL. The aging brain and anesthesia. Curr Opin Anaesthesiol. 2013 Aug;26(4):414-9. doi: 10.1097/ACO.0b013e328362d183. PMID 23820102
- [Background] Monk TG, Weldon BC, Garvan CW, Dede DE, van der Aa MT, Heilman KM, Gravenstein JS. Predictors of cognitive dysfunction after major noncardiac surgery. Anesthesiology. 2008 Jan;108(1):18-30. doi: 10.1097/01.anes.0000296071.19434.1e. PMID 18156878
- [Background] Rudolph JL, Inouye SK, Jones RN, Yang FM, Fong TG, Levkoff SE, Marcantonio ER. Delirium: an independent predictor of functional decline after cardiac surgery. J Am Geriatr Soc. 2010 Apr;58(4):643-9. doi: 10.1111/j.1532-5415.2010.02762.x. Epub 2010 Mar 22. PMID 20345866
- [Background] Jiang L, Hu M, Lu Y, Cao Y, Chang Y, Dai Z. The protective effects of dexmedetomidine on ischemic brain injury: A meta-analysis. J Clin Anesth. 2017 Aug;40:25-32. doi: 10.1016/j.jclinane.2017.04.003. Epub 2017 Apr 17. PMID 28625441
- [Background] Armstrong R, Xu F, Arora A, Rasic N, Syed NI. General anesthetics and cytotoxicity: possible implications for brain health. Drug Chem Toxicol. 2017 Apr;40(2):241-249. doi: 10.1080/01480545.2016.1188306. Epub 2016 Jun 2. PMID 27252089
- [Background] Kant IMJ, de Bresser J, van Montfort SJT, Slooter AJC, Hendrikse J. MRI Markers of Neurodegenerative and Neurovascular Changes in Relation to Postoperative Delirium and Postoperative Cognitive Decline. Am J Geriatr Psychiatry. 2017 Oct;25(10):1048-1061. doi: 10.1016/j.jagp.2017.06.016. Epub 2017 Jun 28. PMID 28760515